CLINICAL TRIAL: NCT01758458
Title: Viral Oncoprotein Targeted Autologous T Cell Therapy for Merkel Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A Phase I/II study (NCT01758458) is now recruiting
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2586.00; NCI-2012-02779 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2586; 2586.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Merkel Cell Carcinoma; Stage IV Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — aldesleukin; Radiotherapy; Radiation; Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (autologous T cells and aldesleukin) (Experimental): Patients undergo radiation therapy or recombinant interferon beta intralesional injection within day -3 to day -1.
  Patients receive MCPyV TAg-specific polyclonal autologous CD8-positive T cell infusion IV on day 1 and aldesleukin SC every 12 hours on days 1-14. Treatment repeats at least every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients with continued presence of detectable metastatic disease 8 weeks after the first infusion may repeat the treatment regimen including radiation therapy or recombinant interferon beta injection.
  Interventions: Biological: Aldesleukin; Other: Laboratory Biomarker Analysis; Biological: MCPyV TAg-specific Polyclonal Autologous CD8-positive T Cells; Radiation: Radiation Therapy; Biological: Recombinant Interferon Beta

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: MCPyV TAg-specific Polyclonal Autologous CD8-positive T Cells — Given IV
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Recombinant Interferon Beta — Given intralesionally
  Other Names: Beta Interferon; Betantrone; Feron; Human Interferon Beta; Interferon Beta; Interferon, Beta; Interferon-B; Interferon-beta; Naferon

SUMMARY:
This phase I/II trial studies the side effects and best way to give laboratory treated autologous T cells together with aldesleukin and to see how well it works in treating patients with merkel cell carcinoma that has spread from the primary site (place where it started) to other places in the body. Biological therapies, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may stimulate the white blood cells to kill tumor cells. Giving cellular adoptive immunotherapy with aldesleukin may be a better treatment for metastatic merkel cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and potential toxicities associated with treating patients with metastatic merkel cell carcinoma (MCC) by combined myosin heavy chain (MHC) up-regulation therapy and adoptive transfer of merkel cell polyomavirus (MCPyV) T-antigen (TAg)-specific polyclonal autologous cluster of differentiation (CD)8+ T cells.

II. Determine the antitumor efficacy associated with treating patients with metastatic MCC by combined MHC up-regulation therapy and adoptive transfer of MCPyV TAg-specific polyclonal autologous CD8+ T cells.

SECONDARY OBJECTIVES:

I. Determine the in vivo persistence and where evaluable, migration to tumor sites of adoptively transferred polyclonal CD8+ T cells targeting the MCPyV TAg.

II. Determine the in vivo functional capacity of adoptively transferred polyclonal CD8+ T cells targeting the MCPyV TAg.

OUTLINE:

Patients undergo radiation therapy or recombinant interferon beta intralesional injection within day -3 to day -1.

Patients receive MCPyV TAg-specific polyclonal autologous CD8-positive T cell vaccine intravenously (IV) on day 1 and aldesleukin subcutaneously (SC) every 12 hours on days 1-14. Treatment repeats at least every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with continued presence of detectable metastatic disease 8 weeks after the first infusion may repeat the treatment regimen including radiation therapy or recombinant interferon beta injection.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological documentation of MCC concurrent with the diagnosis of metastatic disease
* Evidence of MCPyV TAg tumor expression
* Available peptide-MHC pair that can be folded into a tetramer for which MCPyV TAg-specific cells can be generated and reactivity to cell lines expressing MCPyV TAg with the corresponding human leukocyte antigen (HLA)
* Bi-dimensionally measurable disease by palpation, clinical exam, or radiographic imaging (x-ray, computed tomography [CT] scan, positron emission tomography [PET] scan, magnetic resonance imaging [MRI], or ultrasound)
* At least 3 weeks must have passed since any of the following: systemic corticosteroids, immunotherapy (for example, interleukins, MCC vaccines, intravenous immunoglobulin, expanded polyclonal tumor infiltrating lymphocyte [TIL] or lymphokine-activated killer [LAK] therapy), pentoxifylline, other small molecule or chemotherapy cancer treatment, other investigational agents or other agents that target merkel cell carcinoma
* Cardiac ejection fraction >= 40% (multigated acquisition [MUGA] or echocardiogram); for patients with significant risk factors for coronary artery disease (CAD) (including family history, hypertension, and/or dyslipidemia), or age > 50, stress echo or stress thallium testing is required

Exclusion Criteria:

* Unable to generate antigen-specific MCPyV TAg-specific CD8+ T cells for infusions
* Active infections prior to receiving study treatment or systemic infection requiring chronic maintenance or suppressive therapy
* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* White blood cell (WBC) < 2000/mcl
* Hemoglobin (Hb) < 8 g/dL
* Absolute neutrophil count (ANC) < 1000/mcl
* Platelets < 50,000/mcl
* New York Heart Association functional class III-IV heart failure, symptomatic pericardial effusion, stable or unstable angina, symptoms of coronary artery disease, congestive heart failure, clinically significant hypotension, or an ejection fraction of =< 40 % (echocardiogram or MUGA)
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 2.0 L or diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin [Hgb]) < 50% will be excluded
* Creatinine clearance < 30 ml/min which cannot be attributed to MCC metastasis
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN)
* Bilirubin > 3 x ULN which cannot be attributed to MCC metastasis
* Active autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease, inflammatory bowel disease) whose possible progression during treatment would be considered unacceptable by the investigators
* Symptomatic and untreated central nervous system (CNS) metastasis; however, patients with 1-2 asymptomatic, less than 1 cm brain/CNS metastases without significant edema may be considered for treatment; if sub-centimeter CNS lesions are noted at study entry, then a repeat imaging will be performed if more than 4 weeks have elapsed from the last scan
* Any condition or organ toxicity that is deemed by the principal investigator (PI) or the attending physician to place the patient at unacceptable risk for treatment on the protocol
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to entry
* Clinically significant and ongoing immune suppression including, but not limited to, systemic immunosuppressive agents such as cyclosporine or corticosteroids, chronic lymphocytic leukemia (CLL), uncontrolled human immunodeficiency virus (HIV) infection, or solid organ transplantation
* Patients may not be on any other treatments for their cancer aside from those included in the protocol; patients may not undergo another form of treatment concurrently with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Evidence and nature of toxicity related to the study treatment assessed using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4 weeks
  The treatment will be considered to have an acceptable safety profile if the observed toxicity rate is consistent with a true rate that does not exceed 30%.
Evidence of response based on "median time to new metastasis" | Up to 4 years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

SECONDARY OUTCOMES:
Disease response by RECIST criteria | Up to 4 years
Functional capacity of transferred T cells | Up to 4 years
MCC-specific survival | Up to 4 years
Persistence of transferred T cells in blood and in tumor | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chapuis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States